CLINICAL TRIAL: NCT03157648
Title: Relationship Between Core-peripheral Temperature Difference and Shivering Symptom in Patients in PACU
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Other Study IDs: 581/2557
Record Dates: First submitted 2015-07-06; First posted 2017-05-17 (Actual); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Shivering; Body Temperature
Keywords: Shivering temperature

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: observing for shivering symptom — In the PACU investigators measure body temperature of all patients at tympanic membrane, forehead, and dorsal of hand. Investigators calculate the difference between body temperature measure at tympanic membrane and forehead/dorsal of hand. Investigators observe the shivering symptom and grading for severity.

SUMMARY:
Shivering is a physiologic response to early hypothermia in mammals. The definition of shivering is an involuntary, oscillatory muscular activity that augments metabolic heat production.

Routinely in post anesthetic care unit (PACU), the core temperature via tympanic membrane is always measured in all patients. Sometimes patients who have low temperature have no shivering symptom in other hand patients who have normal temperature have shivering symptom. This indicates that, only core temperature is not enough for predicting or detecting patients who will have shivering symptom in PACU.

In this study, investigators hypothesise that the core-peripheral temperature difference in postoperative period indicates patients who will have shivering symptom.

Thus, the aims of this study are to evaluate the relationship between core-peripheral temperature difference and shivering symptom in patients in PACU.

DETAILED DESCRIPTION:
Humans are warm-blooded animal or homeotherms. They are able to regulate their body temperature which in physiologic range themselves. The body temperature is controlled by balancing heat production and heat loss. The normal body temperature refers to either core temperature (eg. tympanic membrane, esophagus, and intra-urinary bladder) or peripheral temperature (eg. skin, forehead, and axillar). Core temperature is the temperature of the deep tissues of the body. The normal range of core temperature is between 36.5-37.5 degree celsius. The peripheral temperature, in contrast to the core temperature, can be changed by many factors such as the temperature of the surroundings environment.

The term of hypothermia is the core temperature less than or equal to 36.4 degree celsius. When the body exposes to cold temperature, heat loss is decreased and heat production is increased as defense mechanism for keeping balance in several means: stop sweating, piloerection, cutaneous arterioles constriction, shivering, which increases heat production in skeletal muscles, conversion from fat to energy by mitochondria.Hypothermia is one of factors, which relates to postoperative complications.

Shivering is an oscillatory muscular activity that augments metabolic heat production. Vigorous shivering increases metabolic heat production up to 600% above basal level. Shivering is a common postoperative period complication. The pathophysiology of postoperative shivering remains unclear otherwise various mechanisms have been proposed. Shivering may happen as a thermoregulatory response to hypothermia or muscle hyperactivity with clonic or tonic patterns. Although cold-induced shivering is an obvious source of postanesthetic tremor. Some of the patients who suffer from shivering are believed to be nonthermoregulatory because their core temperatures remain normal. The incidence of postoperative shivering is 65% of patients after general anesthesia and 33% of patients after regional anesthesia.

This is the prospective observation clinical study. Investigators will observe shivering symptom and measure the patients' temperature at tympanic membrane, forehead, and dorsal of hand at many time points.

ELIGIBILITY:
Inclusion criteria

* Postoperative patient at PACU (Post Anesthesia Care Unit)
* Duration of operation from 1 to 4 hours
* The patients American Society of Anesthesiologist classification from I to III
* The patients' age from 18 years old

Exclusion criteria:

* The patients who reject or unwilling to participate
* The patient who was induced hypothermia in intra-operative period
* The patient who still has neuromuscular blocking agent drugs effect in PACU
* The patient with shock or receiving continuous vasopressor drugs

Withdrawal or termination criteria:

* The patient who has intra-operative or immediate post-operative cardiac arrest and/or death

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who are in the Siriraj PACU at 5th floor Siammintr building. The patients are one of the patients from head-neck-breast surgery, general surgery, or urology surgery.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Difference in temperature | immediate after arriving in PACU
  Difference in temperature measured at tympanic membrane and forehead

SECONDARY OUTCOMES:
Change in temperature | immediate after arriving in PACU
  Difference in temperature measured at tympanic membrane and dorsal hand
Shivering symptom | immediate after arriving in PACU
  Severity of shivering symptom from 0 to 4 grade (0 = No shivering, 1 = No visible muscle activity, but one or more of piloerection, peripheral vasoconstriction or peripheral cyanosis, 2 = Muscular activity in only one muscle group, 3 = Moderate muscular activity in more than one muscle group, but not generalized shaking, 4 = Violent muscular activity that involves the entire body).

CONTACTS AND LOCATIONS:
Overall Officials: Phuriphong Songarj, MD, Principal Investigator — Mahidol University
Locations (1):
- Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Bangkoknoi, Thailand

IPD SHARING:
Plan to Share IPD: No
When the other researcher required data, please direct contact to principle investigator.

REFERENCES:
- See also: Thermoregulation, mild perioperative hypothermia and postanaesthetic shivering. — http://www.ncbi.nlm.nih.gov/pubmed/10844839
- See also: Effects of hypothermia and shivering on standard PACU monitoring of patients. — http://www.ncbi.nlm.nih.gov/pubmed/?term=Effects+of+hypothermia+and+shivering+on+standard+PACU+monitoring+of+patients
- See also: Perioperative shivering: physiology and pharmacology. — http://www.ncbi.nlm.nih.gov/pubmed/?term=Perioperative+Shivering+Physiology+and+Pharmacology
- See also: The intensity of postoperative shivering is unrelated to axillary temperature. — http://www.ncbi.nlm.nih.gov/pubmed/?term=The+intensity+of+postoperative+shivering+is+unrelated+to+axillary+temperature.